CLINICAL TRIAL: NCT00005412
Title: Dietary Antioxidants and Atherosclerosis
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4330; R03HL047408 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2000-06

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Heart Diseases; Carotid Stenosis
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Heart Diseases; Carotid Stenosis

SUMMARY:
To examine the role of dietary antioxidants in the etiology of atherosclerosis in both sexes and in whites and Blacks.

DETAILED DESCRIPTION:
BACKGROUND:

Atherosclerosis is this nation's leading cause of death for males and females, and Blacks and whites. There is mounting evidence that the oxidation of blood low density lipoproteins (LDL) plays an important role in the pathogenesis of this disease. LDL oxidation can be prevented by several dietary antioxidants, in particular, vitamin C, vitamin E, and beta-carotene. There is preliminary evidence that dietary antioxidants may slow the natural history of atherosclerosis in humans. Until now studies in this area have included predominantly white males with symptomatic disease.

DESIGN NARRATIVE:

The case-control study used data collected in ARIC to test the hypothesis that individuals in the lowest quintile of vitamin C, vitamin E and carotenoid consumption were at higher risk of asymptomatic atherosclerosis than those consuming greater amounts. Antioxidant intake was assessed by a validated food frequency questionnaire and a diet supplement survey. Cases were those with asymptomatic carotid artery atherosclerosis as determined by B-mode ultrasonography. Controls were those without evidence of carotid artery atherosclerosis. Secondary analyses determined which sex-race subgroups were at particular risk due to low antioxidant consumption.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1992-07; Study Completion 1995-06 (Actual)

REFERENCES:
- [Background] Kritchevsky SB, Shimakawa T, Tell GS, Dennis B, Carpenter M, Eckfeldt JH, Peacher-Ryan H, Heiss G. Dietary antioxidants and carotid artery wall thickness. The ARIC Study. Atherosclerosis Risk in Communities Study. Circulation. 1995 Oct 15;92(8):2142-50. doi: 10.1161/01.cir.92.8.2142. PMID 7554194
- [Background] Kritchevsky SB, Tell GS, Shimakawa T, Dennis B, Li R, Kohlmeier L, Steere E, Heiss G. Provitamin A carotenoid intake and carotid artery plaques: the Atherosclerosis Risk in Communities Study. Am J Clin Nutr. 1998 Sep;68(3):726-33. doi: 10.1093/ajcn/68.3.726. PMID 9734754